CLINICAL TRIAL: NCT03177642
Title: Orthopaedic Hand and Upper Extremity Data Repository
Status: Withdrawn | Type: Observational
Why Stopped: The data initially planned to be collected under this protocol was transferred into multiple smaller protocols that do not constitute clinical trials. No data was collected under this protocol.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Neal Chung-Jen Chen, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2017P000694
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Non-traumatic and Traumatic Orthopaedic Issues

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Data Repository Group: All adults presenting to the hand and upper extremity service at Massachusetts General Hospital.

SUMMARY:
The purpose of this research is to investigate multiple facets of non-traumatic and traumatic orthopaedic health issues. Studies under this protocol will investigate a variety of research questions concerning traumatic and non-traumatic health issues in the Orthopaedic Hand and Upper Extremity Service.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Patients presenting to the Orthopaedic Hand and Upper Extremity Service for traumatic or non-traumatic issues
* English speaking

Exclusion Criteria:

* Under 18 years
* Vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting to the orthopaedic hand and upper extremity service for a traumatic or non-traumatic issue
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Quick-DASH (Disabilities of the Arm, Shoulder and Hand Quick Questionnaire) | Day 1
  The short form of the Disabilities of Arm Shoulder and Hand to assess upper extremity disability. The scale range is from 0-100, where 0 is no difficulty performing tasks and 100 is the most difficulty or unable to complete any tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No